CLINICAL TRIAL: NCT05970380
Title: Evaluation of the Effect of Erector Spinae Plane Block on Analgesic Consumption in Patients Scheduled for Percutaneous Balloon Kyphoplasty; Prospective Observational Study
Brief Title: Effect of Erector Spinae Plane Block in Patients Scheduled for Kyphoplasty
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halide Hande Şahinkaya, MD, Anesthesiology Specialist, Clinical Director, Bozyaka Training and Research Hospital
Other Study IDs: Kyphoplasty
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Erector Spinae Plane Block
Keywords: percutaneous balloon kyphoplasty; erector spinae plane block; Postoperative Pain; local anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Local

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Local anesthesia: Local anesthesia with 0.25% 20 mL bupivacaine will be given extrapedicular part of the fractured vertebra by the surgeon. At the same time, intravenous 0.1 mg/kg midazolam, 0.3 mg/kg ketamine and 25-100 mcg/kg/min propofol will be administered to achieve sedation and analgesia.
  Interventions: Other: Local anesthesia
- ESP Block: Bilateral erector spinae plane block will be performed at the level of fractured vertebra with totally 40 mL 0.25% bupivacaine under ultrasound imaging by the anesthesiologist. Intravenous 0.1 mg/kg midazolam will be administered for sedation.
  Interventions: Other: Erector spinae plane block

INTERVENTIONS:
Other: Erector spinae plane block — Local anesthetic solution (40 mL 0.25% bupivacaine totally) will be given bilaterally between the processus transversalis of the fractured vertebra and the erector spinae muscle under ultrasound imaging by an anesthesiologist.
  Groups: ESP Block
Other: Local anesthesia — Local anesthetic solution (20 mL 0.25% bupivacaine) will be given extrapedicular part of the fractured vertebra by the surgeon.
  Groups: Local anesthesia

SUMMARY:
Patients, older than 50 years, with vertebral fracture scheduled for percutaneous balloon kyphoplasty will be enrolled for the study. Some patients will be under local anesthesia with sedation and analgesia for the procedure. Some patients will be performed erector spinae plane block with the guidance of ultrasonography for the procedure. The investigators aim to evaluate the intraoperative and postoperative analgesic requirement of patients. Surgeon's and patients' satisfaction will be also evaluated.

DETAILED DESCRIPTION:
Patients, older than 50 years, American Society of Anesthesiologists physical status I, II, III and IV and scheduled for percutaneous balloon kyphoplasty due to osteoporotic vertebra fracture will be enrolled for this prospective, observational study. Written consent will be taken from all patients.

All patients will be taken to the premedication room. Standard monitorization will be performed with electrocardiography, non-invasive blood pressure and pulse oximeter. A 20 Gauge intravenous (iv) canula will be inserted and 10-20 mg/kg iv crystalloid infusion will be started. According to the neurosurgeon's preference patients will be under local anesthesia with sedation and analgesia or erector spinae plane block and sedation during the procedure.

In Group Local Anesthesia (L), local anesthesia with 0.25% 20 mL bupivacaine will be given extrapedicular part of the fractured vertebra by the surgeon. At the same time, intravenous 0.1 mg/kg midazolam, 0.3 mg/kg ketamine and 25-100 mcg/kg/min propofol will be administered to achieve sedation and analgesia.

In Group Erector Spinae Plane Block (ESP), bilateral erector spinae plane block will be performed at the level of fractured vertebra with totally 40 mL 0.25% bupivacaine under ultrasound imaging by the anesthesiologist. 20 minutes after administration of the block, the surgical procedure will be started. During the procedure intravenous 0.1 mg/kg midazolam will be administered for sedation. Pain will be assessed with numeric rating scale (NRS). When NRS is 4 or over 4, additional 0.3 mg/kg ketamine and 25-100 mcg/kg/min propofol will be given intravenously.

In the postoperative period all patients in groups, NRS will be also used to assess the pain. When NRS is 4 or over 4, 1 gr paracetamol will be given intravenously. If NRS will not be under 4 after 1 hour of paracetamol administration, iv 1 mg/kg tramadol will be given.

Postoperative and intraoperative opioid consumption will be assessed to evaluate the effectiveness of erector spinae plane block.

Surgeon's and patients satisfaction will be assessed with 5 points Likert's scale; 1: very dissatisfied, 2: dissatisfied, 3: neither dissatisfied or satisfied, 4: satisfied, 5: very satisfied. All outcome measures will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I, II, III, IV
* Pathologic vertebra fracture
* Percutaneous balloon kyphoplasty for single vertebrae

Exclusion Criteria:

* Contraindications for plane blocks (bleeding disorder, infection on the injection side)
* Hemodynamic instability
* Pregnancy
* Patient's refusal
* Vertebra fracture due to trauma
* Multiple vertebra fractures
* Procedure under general anesthesia
* Allergy to local anesthetics

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologic vertebra fracture that is indicated for percutaneous balloon kyphoplasty will be enrolled for the study.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Opioid consumption during surgery | Within first hour of the surgical procedure
  Opioid consumption will be assessed with the need of opioid analgesics and propofol during the surgical procedure.
Opioid consumption after surgery | Up to 24 hours after the surgical procedure
  Opioid consumption will be assessed with the need of opioid analgesics after the surgery.
Pain during surgical procedure | Within the first hour of the surgical procedure
  Pain during the surgical procedure will be assessed by using numeric rating scale (NRS). NRS is between 0 and 10, where 0 is no pain and 10 is the worst pain. When the NRS is 4 or over 4 additional opioid analgesic will be given to the patient intravenously.
Pain after surgical procedure | Up to 24 hours after the surgical procedure
  Pain will be assessed with numeric rating scale (NRS). NRS is between 0 and 10, where 0 is no pain and 10 is the worst pain. When the NRS is 4 or over 4, additional opioid analgesic will be given to the patient intravenously.

SECONDARY OUTCOMES:
Surgeon's satisfaction | Within 24 hours of the surgical procedure
  The surgeon will assess the ease of the procedure and patient's comfort during the procedure with Likert's scale; 1: very dissatisfied, 2: dissatisfied, 3: neither dissatisfied or satisfied, 4: satisfied, 5: very satisfied
Patient's satisfaction | Within 24 hours of the surgical procedure
  Patient will assess the comfort during intraoperative and postoperative period with Likert's scale 1: very dissatisfied, 2: dissatisfied, 4: neither dissatisfied or satisfied, 4: satisfied, 5: very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Halide H Şahinkaya, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; Alper Tabanlı, MD, Study Chair — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Verduzco LA. Erector spinae plane block as primary anesthetic for kyphoplasty. J Clin Anesth. 2020 May;61:109670. doi: 10.1016/j.jclinane.2019.109670. Epub 2019 Nov 26. No abstract available. PMID 31784307
- [Background] Demir U, Taskin O. Retrospective Comparison of Anesthetic Methods for Percutaneous Balloon Kyphoplasty Surgery: General Anesthesia and Erector Spinae Plane Block. Medicina (Kaunas). 2023 Jan 27;59(2):240. doi: 10.3390/medicina59020240. PMID 36837442
- [Background] Ge C, Wu X, Gao Z, Xu Z, Hao D, Dong L. Comparison of different anesthesia modalities during percutaneous kyphoplasty of osteoporotic vertebral compression fractures. Sci Rep. 2021 May 27;11(1):11102. doi: 10.1038/s41598-021-90621-9. PMID 34045557
- [Background] Wu AM, Lin ZK, Ni WF, Chi YL, Xu HZ, Wang XY, Huang QS. The existence of intravertebral cleft impact on outcomes of nonacute osteoporotic vertebral compression fractures patients treated by percutaneous kyphoplasty: a comparative study. J Spinal Disord Tech. 2014 May;27(3):E88-93. doi: 10.1097/BSD.0b013e31829142bf. PMID 23563348